CLINICAL TRIAL: NCT03702127
Title: Investigating the Effects of Transcranial Magnetic Stimulation With Intracranial EEG in Humans
Brief Title: TMS - Intracranial Electrodes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aaron Boes (Other)
Collaborators: Stanford University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Aaron Boes, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201707763; 1R21MH120441-01 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Masking Description: Participant will receive active and sham stimulation at varying points during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMS in patients with intracranial electrodes (Experimental): We will administer TMS to neurosurgical patients with intracranial electroencephalography in order to better understand the effects TMS has on the human brain. Participants will receive both active and sham stimulation at varying points during the study.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — NIBS is applied to the brain.

SUMMARY:
This is a study looking at the effects of transcranial magnetic stimulation (TMS), a form of non-invasive brain stimulation (NIBS), on the human brain as recorded by intracranial electroencephalography in neurosurgical patients. NIBS will be applied in a targeted manner and brain responses will be recorded.

DETAILED DESCRIPTION:
In the last few years, non-invasive brain stimulation techniques such as transcranial magnetic stimulation (TMS), transcranial current stimulation, and peripheral multi-modal stimulation have shown widespread clinical applications. Transcranial magnetic stimulation (TMS) is a noninvasive method of focally stimulating the brain that uses electromagnetic induction and does not require surgery. There is optimism that TMS and other forms of NIBS will revolutionize how we treat neurological and psychiatric disorders, evidenced by over 1000 clinical trials registered using TMS. Much of this optimism stems from the successful use of TMS as a treatment for depression. Despite the large number of clinical trials using NIBS the number of therapeutic indications has been stagnant, limited to major depression and more recently obsessive-compulsive disorder. There are fundamental questions about the underlying mechanisms of action for NIBS that will be critical to understand in order to advance this treatment modality. Here, we propose a unique collaborative project between neurology and neurosurgery that will allow an unprecedented window into understanding how NIBS impacts the human brain. Specifically, we will perform various forms of targeted TMS in neurosurgical patients with intracranial electroencephalography (iEEG) monitoring to record real time effects of NIBS on local and remote brain areas with an unparalleled combination of spatial and temporal resolution relative to other human studies. TMS may present the most risk for patients with intracranial electrodes and we have already demonstrated the safety of this approach using a gel-based phantom brain and have results from seven patients demonstrating safety and preliminary results. For the current proposal we aim to: 1) characterize the response of NIBS on the human brain as recorded from iEEG between active and sham conditions, and 2) relate remote electrophysiological responses from NIBS to measures of brain connectivity between the stimulation & recording sites assessed with resting state functional connectivity MRI (rs-fcMRI). This will allow us to evaluate the relationship between NIBS-evoked iEEG responses and the strength of functional connectivity to the stimulation site in a regression model. For the TMS portion of the study we hypothesize that 1) TMS will have focal effects detected from surface electrodes underlying the stimulation site as well as network-level engagement detected at remote sites, 2) Repetitive TMS will induce frequency-specific effects that differ between 0.5 and 10 Hz stimulation protocols, and 3) the magnitude of repetitive TMS-evoked iEEG responses across electrodes will relate to the strength of rs-fcMRI between the stimulation and recording sites. By investigating the electrophysiological responses of TMS with high spatiotemporal precision in humans, this study will provide new mechanistic insights into the effects of TMS on target engagement and relate these findings to imaging methods already in widespread use. Moreover, the TMS will be applied in a clinically meaningful way by targeting the left dorsolateral prefrontal cortex in a protocol used to treat depression. Generating results for these aims will be key to advancing our understanding of how TMS and other forms of NIBS engage brain networks, which can be leveraged to rationally develop personalized, imaging-guided therapeutic NIBS for depression and other disorders.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will include neurosurgery patients (age 18 and above) who have implantation of intracranial electrodes and undergo long term (about 2 weeks) EEG monitoring in order to decide candidacy for surgical resection of seizure foci. They must have the cognitive capacity to understand the risks and benefits fo the study and provide consent.

Exclusion Criteria:

Those who are known to have neurological or psychiatric disorder other than primary disease for which patients have surgery will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity assessed with intracranial EEG | Activity changes within seconds of the stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Boes, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No